CLINICAL TRIAL: NCT03883113
Title: Efficacy of MVA-NP+M1 in the Influenza H3N2 Human Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barinthus Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLU010
Record Dates: First submitted 2019-02-21; First posted 2019-03-20 (Actual); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MVA-NP+M1 & H3N2 Challenge Virus (Experimental): Vaccination administered: MVA-NP+M1 (IM injection, 0.5 ml, 1.5 x10^8 pfu.); Challenge Virus administered: H3N2 (nasal spray, 0.5 ml, 1.0x10^6 TCID50/ml)
  Interventions: Biological: MVA-NP+M1; Biological: H3N2 (A/Belgium/2417/2015)
- Saline Placebo & H3N2 Challenge Virus (Placebo Comparator): Vaccination administered: Sodium Chloride (IM injection, 0.5 ml, 0.9%); Challenge Virus administered: H3N2 (nasal spray, 0.5 ml, 1.0x10^6 TCID50/ml)
  Interventions: Biological: Saline; Biological: H3N2 (A/Belgium/2417/2015)

INTERVENTIONS:
Biological: MVA-NP+M1 — Trial Vaccine
  Arms: MVA-NP+M1 & H3N2 Challenge Virus
Biological: Saline — Sodium Chloride Placebo
  Arms: Saline Placebo & H3N2 Challenge Virus
Biological: H3N2 (A/Belgium/2417/2015) — Challenge Agent

SUMMARY:
A Phase 2, single center, randomized, double blind study evaluating the safety, efficacy, and immunogenicity of MVA NP+M1 in the H3N2 human influenza challenge model; on healthy adult volunteers.

DETAILED DESCRIPTION:
The study consists of an outpatient vaccination phase (155 participants), and at least 2 months later an inpatient challenge phase (134 participants). Participants are randomized 93:62 to receive either MVA-NP+M1 or Placebo. Up to 20 participants will be challenged over several 3-week blocks, and the remainder at the final 3-week block for a total of 80 MVA-NP+M1 and 54 Placebo recipients challenged.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged ≥18 and ≤55 years of age at the point of enrolment.
* Non-smokers or those who stopped smoking ≥ 3 months prior to screening 1 visit.
* Willingness to remain in isolation for the duration of the study.
* A female participant is eligible for this study if she is not pregnant or breast feeding and 1 of the following:

  1. Of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
  2. Of childbearing potential but has been and agrees to continue practicing highly effective contraception or abstinence (if this is the preferred and usual lifestyle of the participant) from 6 months prior to vaccination to 6 months after administration of the influenza challenge virus. Highly effective methods of contraception include 1 or more of the following:

  i. male partner who is sterile (vasectomised) prior to the female participants entry into the study and is the sole sexual partner for the female participant; ii. hormonal (oral, intravaginal, transdermal, implantable or injectable); iii. an intrauterine hormone-releasing system (IUS); iv. an intrauterine device (IUD) with a documented failure rate of < 1%; v. bilateral tubal occlusion.
* Pre-challenge serum microneutralization test (MNT) against A/Belgium/4217/2015 (H3N2) challenge strain < 20.

Exclusion Criteria:

* BMI < 19 and > 32.
* Presence of any significant acute or chronic, uncontrolled medical (or psychiatric) illness including a history of chronic respiratory illness.
* History of seasonal hay fever or a clinically significant seasonal allergic rhinitis (SAR), including the use of symptomatic prescription only medication and non-prescription medication.
* History or evidence of autoimmune disease or known immunodeficiency of any cause - with the exception of atopic dermatitis/eczema and atopic rhinitis.
* Any history of anaphylaxis in reaction to vaccination or history of allergic reactions likely to be exacerbated by any component of the vaccine.
* History of lung disease (Asthma, COPD).
* Current smokers or those who stopped smoking < 3months prior to screening 1 visit.
* Positive diagnostic tests for HIV, Hepatitis B or Hepatitis C indicating active infection.
* Evidence of drug abuse or a positive urine drug screen or alcohol breath test.
* Chronic use of any medication or other product (prescription or over-the-counter), for symptoms of rhinitis or nasal congestion or for any chronic nasopharyngeal complaint, or chronic use of any intranasal medication for any indication that has not ceased within 30 days prior to screening 1.
* Receipt of any investigational drug within 3 months prior to vaccination, or prior participation in a clinical trial of any influenza vaccine, or any investigational vaccine or experimental influenza viral challenge delivered directly to the respiratory tract within 1 year prior to challenge.
* Receipt of the 2018/2019 seasonal flu vaccine.
* Receipt of any live vaccines within the 4 weeks prior to vaccination.
* Any laboratory test which is abnormal and which is deemed by the Investigator(s) to be clinically significant.
* Receipt of any systemic chemotherapy agent at any time.
* Physician reported influenza or a syndrome consistent with influenza (as judged by the investigator) in the previous 6 months.
* Known allergy to treatments for influenza (including but not limited to oseltamivir).
* History of frequent epistaxis (nose bleeds).
* Any nasal or sinus surgery within 6 months of Viral Challenge or any significant abnormality, either of which results in alteration of the anatomy of the nose or nasopharynx (including significant nasal polyps).
* Volunteers with household contacts who are at risk for serious or severe complications of influenza disease including, but not limited to: persons ≥ 65 years; presence of significant chronic cardiopulmonary, metabolic, renal, or neurological conditions; immunosuppression due to any condition or therapies; BMI >40.
* Participants that are an employee or family member of the Investigator or study site personnel may not be enrolled.
* Any other finding that, in the opinion of the Investigator, deems the participant unsuitable for the study.

EXCLUSION (CHALLENGE PERIOD ONLY)

* Abnormal spirometry assessed to be clinically significant.
* Known close contact with anyone known to have influenza in the past 7 days at the time of quarantine.
* Influenza-like illness (ILI) symptoms as assessed at the admission to clinic on Day -2 prior to challenge.
* Presence of fever, defined as participant presenting with a temperature reading of > 38.0°C on admission to quarantine.
* Qualitative Polymerase chain reaction (PCR) results positive for viral infection. However, participants may be included into later challenge cohort.
* Acute use of any medication or other product, prescription or over-the-counter, for symptoms of rhinitis or nasal congestion within 7 days prior to challenge. This includes any oral corticosteroid or beta agonist containing nasal spray.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Rogiers, MD, Principal Investigator — SGS S.A.
Locations (1):
- SGS Life Sciences, Clinical Pharmacology Unit (CPU), Antwerp, Belgium

REFERENCES:
- [Derived] Evans TG, Castellino F, Kowalik Dobczyk M, Tucker G, Walley AM, Van Leuven K, Klein J, Rutkowski K, Ellis C, Eagling-Vose E, Treanor J, van Baalen C, Filkov E, Laurent C, Thacker J, Asher J, Donabedian A. Assessment of CD8+ T-cell mediated immunity in an influenza A(H3N2) human challenge model in Belgium: a single centre, randomised, double-blind phase 2 study. Lancet Microbe. 2024 Jul;5(7):645-654. doi: 10.1016/S2666-5247(24)00024-7. Epub 2024 May 7. PMID 38729196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the SGS Clinical Pharmacology Unit in Antwerp, Belgium.
Pre-assignment Details: Eight-hundred and nineteen (819) subjects were screened. One hundred and forty-five (145) subjects were actually enrolled and vaccinated. The study consisted of an outpatient vaccination phase and at least 6 weeks later an inpatient challenge phase.
Period: Overall Study
Arm/Group | MVA-NP+M1 & H3N2 Challenge Virus | Saline Placebo & H3N2 Challenge Virus
Started | 87 | 58
Completed | 71 | 46
Not Completed | 16 | 12
Not completed — Physician Decision | 4 | 2
Not completed — Challenge Criteria Not Met / Sponsor Decision | 9 | 7
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVA-NP+M1 & H3N2 Challenge Virus | Saline Placebo & H3N2 Challenge Virus | Total
Number analyzed (Participants) | 87 | 58 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 58 | 145
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 43.00 [18.5 to 55.9] | 41.25 [19.9 to 55.7] | 42.50 [18.5 to 55.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 31 | 78
  Male | 40 | 27 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black or African American | 4 | 0 | 4
  Middle Eastern | 0 | 1 | 1
  White | 81 | 57 | 138
Region of Enrollment [Number; unit: participants]
  Belgium | 87 | 58 | 145
Smoking Status [Count of Participants; unit: Participants]
  Ex-smoker | 27 | 18 | 45
  Non-smoker | 60 | 40 | 100
Height [Median (Full Range); unit: cm] | 172.40 [153.2 to 193.3] | 172.30 [151.8 to 191.7] | 172.40 [151.8 to 193.3]
Weight [Median (Full Range); unit: kg] | 72.9 [53.2 to 118.8] | 75.15 [54.6 to 105.6] | 73.60 [53.2 to 118.8]
BMI [Median (Full Range); unit: kg/m^2] | 24.7 [19.0 to 32] | 25.5 [19.2 to 31.2] | 24.90 [19.0 to 32.0]

OUTCOME MEASURES:

1. Primary Outcome: Degree of Nasopharyngeal Viral Shedding as Determined by Quantitative Polymerase Chain Reaction qPCR
Description: Measure of nasopharyngeal viral shedding during challenge; recorded as viral area under curve (vAUC) as determined by quantitative real time polymerase chain reaction (qRT-PCR). vAUC is calculated by plotting the log viral particles number/ml for each time point against time and is using the trapezoidal rule.
Time Frame: Throughout 9 days (Day2, Day3, Day4, Day5, Day6, Day7, Day8, Day9, Day10) after viral Inoculation (Day1) of the challenge phase. Nasal swabs taken twice a day (b.i.d) at least 8 hours apart.
Population: End point values
Measure: Least Squares Mean (95% Confidence Interval); unit: hour*Log10 Viral Particles/ ml
Groups:
- MVA-NP+M1 (ITT); Placebo (ITT): Intention-to-treat (the actually challenged with the virus)
- MVA-NP+M1 (PP); Placebo (PP): Per protocol analysis set
- MVA-NP+M1 (Challenge); Placebo (Challenge): Safety Analysis Set (challenged participants)
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT) | MVA-NP+M1 (PP) | Placebo (PP) | MVA-NP+M1 (Challenge) | Placebo (Challenge)
Number analyzed (Participants) | 71 | 47 | 70 | 47 | 71 | 47
hour*Log10 Viral Particles/ ml | 649.7 [552.7 to 746.7] | 726.1 [604.0 to 848.2] | 646.5 [548.3 to 744.7] | 726.1 [604.0 to 848.2] | 649.7 [552.7 to 746.7] | 726.1 [604.0 to 848.2]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); Test type: Other; p = 0.1711, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: MVA-NP+M1 (PP) vs Placebo (PP); Test type: Other; p = 0.1654, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: MVA-NP+M1 (Challenge) vs Placebo (Challenge); Test type: Other; p = 0.1711, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number and Percentage of Virologically Confirmed Influenza-Like Illness
Description: Incidence (frequency tabulation) of laboratory-confirmed influenza-like illness compared between vaccine and placebo arms Virologically confirmed influenza-like illness (ILI) is defined as having respiratory or flu-like symptom occurring on two consecutive days, along with a positive qPCR or qCulture result.
Time Frame: 9 days from day 2 to day 10
Measure: Count of Participants; unit: Participants
Groups:
- MVA-NP+M1 (ITT); Placebo (ITT): Intention-to-treat
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
Participants
  Virologically confirmed Influenza-like Illness | 43 | 29
  No Virologically Confirmed Influenza-like Illness | 28 | 18
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); The statistical analysis applies to participants with Virologically confirmed Influenza-like Illness versus participants without Virologically confirmed Influenza-like Illness; Test type: Other; p = 1.000, Fisher Exact

3. Secondary Outcome: Percentage of Participants With Attack Rate of Challenge Agent (qRT-PCR)
Description: The attack rate is defined as the percentage of inoculated participants with at least two consecutive positive swabs as determined by qRT-PCR within the timespan of two consecutive days
Time Frame: 9 days from day 2 to day 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
percentage of participants
  qPCR-confirmed influenza | 90.1 [80.7 to 95.9] | 97.9 [88.7 to 99.9]
  No qPCR influenza | 9.9 [4.1 to 19.3] | 2.1 [0.1 to 11.3]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); This statistical analysis applies to participants with qPCR confirmed Influenza versus participants with no qPCR confirmed Influenza; Test type: Other; p = 0.143, Fisher Exact

4. Secondary Outcome: Percentage of Participants With Quantitative Culture Attack Rate of Challenge Agent (qCulture)
Description: The attack rate is defined as the percentage of inoculated participants with at least two consecutive positive swabs as determined by qCulture within the timespan of two consecutive days
Time Frame: 9 days from day 2 to day 10
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
percentage
  qCulture confirmed influenza | 77.5 [66.0 to 86.5] | 85.1 [71.7 to 93.8]
  No qCulture-confirmed influenza | 22.5 [13.5 to 34.0] | 14.9 [6.2 to 28.3]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); This statistical analysis applies to participants with qCulture confirmed Influenza versus participants without qCulture confirmed Influenza; Test type: Other; p = 0.3504, Fisher Exact

5. Secondary Outcome: Time to Start of Viral Shedding (qPCR) From Virus Inoculation
Description: The Time to Start of Viral Shedding (qPCR) is calculated as (datetime of first of two positive swabs (qPCR) within 2 consecutive days - challenge datetime)/(60*60)
Time Frame: 9 days from day 2 to day 10
Population: [MVA-NP+M1 (ITT)] - subjects assessed = 71 subjects with event = 64 subjects censored = 7 [Placebo (ITT)] - subjects assessed = 47 subjects with event = 46 subjects censored = 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
hours | 24.40 [24.30 to 24.50] | 24.30 [24.20 to 24.50]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); Test type: Other; p = 0.5558, Log Rank

6. Secondary Outcome: Time to Start of Viral Shedding (qCulture) From Virus Inoculation
Description: Time to Start of Viral Shedding (qCulture) is calculated as (datetime of first of two positive swabs (qCulture) within 2 consecutive days - challenge datetime)/(60*60)
Time Frame: 9 days from day 2 to day 10
Population: [MVA-NP+M1(ITT)] - Subjects assessed = 71 Subjects with event = 55 Subjects censored = 16; [Placebo (ITT)] - Subjects assessed = 47 Subjects with event = 40 Subjects censored = 7
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
hours | 35.9 [35.60 to 48.00] | 47.6 [24.70 to 48.50]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); Test type: Other; p = 0.6534, Log Rank

7. Secondary Outcome: Peak Viral Shedding (qPCR) After the Virus Inoculation
Description: This is measured by the highest viral load concentration by qPCR
Time Frame: 9 days from Day 2 to Day 10
Measure: Mean (95% Confidence Interval); unit: Log10 Viral Particles/ ml
Groups:
- MVA-NP+M1 (ITT) Successful Attack: Subset of participants who received MVA-NP+M1 and with a successful attack
- Placebo (ITT) Successful Attack: Subset of participants who received Placebo and with a successful attack
Arm/Group | MVA-NP+M1 (ITT) Successful Attack | Placebo (ITT) Successful Attack
Number analyzed (Participants) | 64 | 46
Log10 Viral Particles/ ml | 5.876 [5.430 to 6.322] | 6.054 [5.521 to 6.587]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) Successful Attack vs Placebo (ITT) Successful Attack; Test type: Other; p = 0.5485, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Peak Viral Shedding (qCulture) After Virus Inoculation
Description: This is measured by the highest viral load concentration by qCulture.
Time Frame: 9 days from day 2 to day 10
Measure: Mean (95% Confidence Interval); unit: Log10 Viral Particles/ ml
Arm/Group | MVA-NP+M1 (ITT) Successful Attack | Placebo (ITT) Successful Attack
Number analyzed (Participants) | 55 | 40
Log10 Viral Particles/ ml | 4.073 [3.683 to 4.463] | 4.069 [3.442 to 4.695]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) Successful Attack vs Placebo (ITT) Successful Attack; Test type: Other; p = 0.6753, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Time to Peak of Viral Shedding (qPCR) From the Viral Inoculation
Description: This is calculated as (datetime of highest viral load concentration (qPCR) - challenge datetime)/(60*60)
Time Frame: 9 days from day 2 to day 10
Population: [MVA-NP+M1 (ITT)] - Subjects assessed = 71 Subjects with event = 64 Subjects censored = 7; [Placebo (ITT)] - Subjects assessed = 47 Subjects with event = 46 Subjects censored = 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
hours | 72.20 [60.00 to 96.00] | 107.90 [72.20 to 119.80]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); Test type: Other; p = 0.711, Log Rank

10. Secondary Outcome: Time to Peak of Viral Shedding (qCulture) From the Viral Inoculation
Description: This is calculated as (datetime of highest viral load concentration (qCulture) - challenge datetime)/(60*60)
Time Frame: 9 days from day 2 to day 10
Population: [MVA-NP+M1 (ITT)] - Subjects assessed = 71 Subjects with event = 55 Subjects censored = 16; [Placebo (ITT)] - Subjects assessed = 47 Subjects with event = 40 Subjects censored = 7
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
hours | 83.40 [60.10 to 96.30] | 83.80 [60.10 to 96.40]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); Test type: Other; p = 0.4689, Log Rank

11. Secondary Outcome: Duration of Viral Shedding (qPCR) After the Virus Inoculation
Description: It is calculated as (datetime of first negative swab (qPCR) following the last positive swab (qPCR) - datetime of first positive of two positive swabs (qPCR) within 2 consecutive days)/(60*60)
Time Frame: 9 days from day2 to day10
Population: This endpoint is only calculated for the subset of participants with a successful attack.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | MVA-NP+M1 (ITT) Successful Attack | Placebo (ITT) Successful Attack
Number analyzed (Participants) | 64 | 46
hours | 170.80 [157.08 to 184.52] | 172.47 [156.99 to 187.94]

12. Secondary Outcome: Duration of Viral Shedding (qCulture) After the Virus Inoculation
Description: It is calculated as (datetime of first negative swab (qCulture) following the last positive swab (qCulture) - datetime of first positive of two positive swabs (qCulture) within 2 consecutive days)/(60*60)
Time Frame: 9 days from day 2 to day 10
Population: This endpoint is only calculated for the subset of participants with a successful attack
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | MVA-NP+M1 (ITT) Successful Attack | Placebo (ITT) Successful Attack
Number analyzed (Participants) | 55 | 40
hours | 118.19 [105.07 to 131.31] | 121.78 [106.33 to 137.23]

13. Secondary Outcome: Total Area Under the Curve (AUC) of Self-reported Influenza Total Symptom Score (SSC AUC)
Description: Total symptom scores were compared for MVA-NP+M1 vs. Placebo from Day1 to Day11 post-challenge as AUC of composite score.
  Symptoms were collected twice a day (lymphadenopathy once a day) on a Symptom Score Card(SSC).
  SSC recorded scores for each 16 general (gastrointestinal/body systemic) and 12 local (upper/lower respiratory tract) symptoms, on the scale per timepoint (for example Day2,AM).
  Participants rated the severity of symptoms, higher scores indicating a more severe symptom.
  The scores ranged from 0 to 3 (0:symptom free, 1:mild, 2:moderate, 3:severe).The SSC also contained the question whether the subject felt well to go to work "today" (yes/no). The Overall SSC score was calculated, as the Arithmetic Mean of the Scores collected across all 28 items on the card per Timepoint and ranged from 0 to maximum 3.
  The SSC AUC [0-11 days] was derived based on the Overall SSC score against time (*hour), using the linear trapezoidal rule and it ranged from 0 to 110 Score*hour.
Time Frame: 11 days from Day 1 to Day 11
Measure: Geometric Mean (95% Confidence Interval); unit: Composite symptom score on scale*hour
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
Composite symptom score on scale*hour | 16.709 [11.568 to 21.850] | 20.432 [13.753 to 27.112]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); Test type: Other; p = 0.5001, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Total Days of Fever
Description: Total days of fever for MVA-NP+M1 vs. Placebo
Time Frame: 11 days from Day 1 to Day 11
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
days | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); Test type: Other; p = 0.6799, zero-inflated poisson model

15. Secondary Outcome: Average Total Mucus Production
Description: Total mucus weight of used tissue (regardless of take rate) for MVA-NP+M1 vs. Placebo.
  Total mucus production was only be calculated in case all tissues were returned (sum of clean and used tissues returned should be 20 tissues for each bag).
Time Frame: 11 days from Day 1 to Day 11
Population: Total mucus production was only calculated for challenge cohorts 5 to 8 and only if all tissues (cleaned or used) were returned.
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 26 | 18
grams | 31.09 [16.23 to 45.85] | 38.21 [16.78 to 59.63]
Statistical Analysis 1: Comparison: MVA-NP+M1 (ITT) vs Placebo (ITT); Test type: Other; p = 0.5911, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: T Cell Responses as Defined by ELISpot Assay in Relation to the Primary Endpoint, Symptom Scores and Influenza Incidence
Description: T Cell Response was assessed for IFN gamma and granzyme B, on the peripheral blood mononuclear cell using a double-colour enzymatic ELISpot assay.
  For each of them, three stimulation antigens were assessed: nucleoprotein NP, matrix1 M1 and a negative control, dimethyl sulfoxide (DMSO).
  The number of spot-forming T cell colonies per well (i.e. 200,000 cells) +/- standard deviation for the total response to NP+M1 is reported.
  The endpoint was recorded as the mean spot-forming units per million peripheral blood mononuclear cells in the peptide-stimulated wells minus the mean DMSO control wells for the sample. T cell responses over time (sampling timepoints) were then assessed in relation to the primary endpoint, symptom scores, and influenza incidence.
Time Frame: 3 months (day 0, day 8 and day 28 of the vaccination period and day -1 and day 28 of the challenge period)
Measure: Mean (Standard Deviation); unit: Spot-forming units per million
Arm/Group | MVA-NP+M1 (ITT) | Placebo (ITT)
Number analyzed (Participants) | 71 | 47
Spot-forming units per million
  Baseline (Vaccination) | 230 (265) | 167 (157)
  Day 8 (from Vaccination) | 645 (634) | 170 (144)
  Day 28 (from Vaccination) | 566 (551) | 163 (160)
  Day 0 Challenge Period | 460 (471) | 159 (132)
  Day 28 Challenge Period | 561 (483) | 329 (220)

17. Secondary Outcome: Number of Participants With MVA-NP+M1 Vaccination Related Adverse Events and Symptoms, Measured by Self-reported Symptoms
Description: Occurrence of solicited local and systemic reactogenicity signs and symptoms for 7 days following vaccination; self-reported symptoms recorded using paper diaries
Time Frame: 7 days following vaccination
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- MVA-NP+M1: Vaccination administered: MVA-NP+M1 (IM injection, 0.5 ml, 1.5 x10^8 pfu.); Challenge Virus administered: H3N2 (nasal spray, 0.5 ml, 1.0x10^6 TCID50/ml)
  MVA-NP+M1: Trial Vaccine
- Saline Placebo: Vaccination administered: Sodium Chloride (IM injection, 0.5 ml, 0.9%); Challenge Virus administered: H3N2 (nasal spray, 0.5 ml, 1.0x10^6 TCID50/ml)
  Saline: Sodium Chloride Placebo
Arm/Group | MVA-NP+M1 | Saline Placebo
Number analyzed (Participants) | 87 | 58
Participants
  TEAE | 36 | 18
  Solicited symptom | 84 | 24
  TEAE or solicited symptom | 85 | 34
  Local solicited symptom | 80 | 8
  Local Grade 3 solicited symptom | 2 | 0
  Systemic solicited symptom | 72 | 20
  Systemic Grade 3 solicited symptom | 2 | 0
  TEAE of special interest | 0 | 0
  Serious TEAE | 1 | 0
  Non-serious TEAE | 36 | 18
  Grade ≥3 TEAE | 1 | 0
  Grade ≥3 TE laboratory toxicity | 2 | 0
  Fatal TEAE | 0 | 0
  TEAE related to treatment | 10 | 4
  Serious TEAE related to treatment | 1 | 0
  Grade ≥3 TEAE related to treatment | 1 | 0
  TEAE for which the study was discontinued | 0 | 0

18. Secondary Outcome: Number of Participants With H3N2 Challenge Related Adverse Events and Symptoms, Measured by Self-reported Symptoms
Description: Occurrence of solicited local and systemic reactogenicity signs and symptoms; self-reported symptoms recorded using questionnaires and adverse event monitoring
Time Frame: 17 days following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-NP+M1 (Challenge) | Placebo (Challenge)
Number analyzed (Participants) | 71 | 47
Participants
  TEAE | 30 | 21
  Solicited symptom | 62 | 40
  TEAE or solicited symptom | 65 | 42
  Local solicited symptom | 59 | 39
  Local Grade 3 solicited symptom | 0 | 0
  Systemic solicited symptom | 45 | 32
  Systemic Grade 3 solicited symptom | 0 | 0
  TEAE of special interest | 0 | 0
  Serious TEAE | 0 | 1
  Non-serious TEAE | 30 | 20
  Grade ≥3 TEAE | 0 | 2
  Grade ≥3 TE laboratory toxicity | 7 | 2
  Fatal TEAE | 0 | 0
  TEAE related to challenge | 7 | 5
  Serious TEAE related to challenge | 0 | 0
  Grade ≥3 TEAE related to challenge | 0 | 0
  TEAE for which the study was discontinued | 0 | 1

19. Other Pre Specified Outcome: Severity of Individual Symptoms for MVA-NP+M1 vs. Placebo
Description: Severity of individual self-reported symptoms for MVA-NP+M1 vs. Placebo
Time Frame: 11 days
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Total Symptom Score Time to Start, Time to Peak and Duration
Description: Time to start; time to peak and duration of total self-reported symptom score, regardless of take rate
  Influenza Symptom Score Card of FLU010 - Solicited symptoms for generalized, and upper and lower respiratory tract symptoms scored by severity (0: absent, 1: mild, 2: moderate, or 3: severe).
Time Frame: 11 days
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Correlation of T Cell Phenotypes With Illness Outcomes
Description: Correlation of antigen specific T Cell phenotypes with illness outcomes
Time Frame: 3 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Vaccination Effect on Antibody Responses by ELISpot and ICS Assays
Description: Antibody responses of MVA-NP+M1 vs Placebo following influenza challenge measured by ELISpot and Intracellular Cytokine Staining (ICS)
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Any time during the study from the first administration of any study drug until the last study-related activity (the outpatient visit at 27 days ±3 days following the challenge or 6 months following vaccination ±14 days, whichever is longer)
Description: Treatment-emergent adverse events (TEAE) are defined as the Adverse Events starting during or after first administration of any study drug to the end of the study independently of their intensity and if they are related or not to the study drug.
Groups:
- MVA-NP+M1 (Vaccination Phase): Vaccination administered: MVA-NP+M1 (IM injection, 0.5 ml, 1.5 x10^8 pfu.);
  MVA-NP+M1: Trial Vaccine
- Saline Placebo (Vaccination Phase): Vaccination administered: Sodium Chloride (IM injection, 0.5 ml, 0.9%);
  Saline: Sodium Chloride Placebo
- MVA-NP+M1 (Challenge Phase): Vaccination administered: MVA-NP+M1 (IM injection, 0.5 ml, 1.5 x10^8 pfu.);
  MVA-NP+M1: Trial Vaccine
  Challenge Virus administered: H3N2 (nasal spray, 0.5 ml, 1.0x10^6 TCID50/ml)
- Saline Placebo (Challenge Phase): Vaccination administered: Sodium Chloride (IM injection, 0.5 ml, 0.9%);
  Saline: Sodium Chloride Placebo
  Challenge Virus administered: H3N2 (nasal spray, 0.5 ml, 1.0x10^6 TCID50/ml)
Arm/Group | MVA-NP+M1 (Vaccination Phase) | Saline Placebo (Vaccination Phase) | MVA-NP+M1 (Challenge Phase) | Saline Placebo (Challenge Phase)
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/58 | 0/71 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/87 | 0/58 | 0/71 | 1/47
Other Adverse Events (participants affected / at risk) | 36/87 | 18/58 | 30/71 | 21/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVA-NP+M1 (Vaccination Phase) (N=87) | Saline Placebo (Vaccination Phase) (N=58) | MVA-NP+M1 (Challenge Phase) (N=71) | Saline Placebo (Challenge Phase) (N=47)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVA-NP+M1 (Vaccination Phase) (N=87) | Saline Placebo (Vaccination Phase) (N=58) | MVA-NP+M1 (Challenge Phase) (N=71) | Saline Placebo (Challenge Phase) (N=47)
Nasopharyngitis (Infections and infestations) | 6 (7) | 4 (4) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 3 (3) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 2 (2) | 1 (1)
Dizziness Postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 4 (4) | 6 (6)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation Increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling of Eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Scar Excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03883113/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT03883113/SAP_001.pdf